CLINICAL TRIAL: NCT05877001
Title: An Open Label, Single-center Study on the Safety of Hepatic Arterial Infusion Chemotherapy Combined With Tislelizumab and Regorafenib in Patients With Advanced Treated Colorectal Liver Metastases
Brief Title: The Safety and Efficacy of HAIC+Tislelizumab+Regorafenib in Patients With Colorectal Liver Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022KT98
Record Dates: First submitted 2023-01-17; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2022-12

CONDITIONS: Colorectal Liver Metastases
MeSH Terms: interventions — tislelizumab; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAIC combined with Tislelizumab and Regorafenib (Experimental): HAIC combined with Tislelizumab and Regorafenib until progression or death.
  Interventions: Drug: Tislelizumab; Drug: Regorafenib; Other: HAIC

INTERVENTIONS:
Drug: Tislelizumab — 200mg, IV, Q3W
  Other Names: BGB-A317
Drug: Regorafenib — 80 mg once daily for the first 3 weeks of each 4-week cycle
  Other Names: BAY73-4506
Other: HAIC — OXA 85mg/m2 IA 0-4h +5-Fu 2000mg/m2 IA 4-48h，CF 200mg/m2 IV 2-4h， Q3W

SUMMARY:
Tislelizumab is an anti-PD-1 monoclonal antibody with high binding affinity for PD-1 and with minimized Fcγ receptor binding on macrophages. Regorafenib has been approved in mCRC by CFDA. Hepatic arterial infusion chemotherapy has a high local control rate for liver metastases. NCCN guidelines and several expert consensus recommend that regional hepatic arterial infusion chemotherapy can be considered as a "rescue treatment" for patients with colorectal cancer liver metastases who fail to receive first-line or second-line systemic chemotherapy, which can significantly prolong the overall survival of patients.

DETAILED DESCRIPTION:
The investigators aimed to evaluated the safety and efficacy of HAIC combined with Tislelizumab and Regorafenib in patients with advanced treated colorectal liver metastases. This study is a prospective, open label, single-center clinical study and the sample size is 20.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years old
2. Histologically or cytologically confirmed colorectal cancer with unresectable or surgical contraindicated liver metastases

   * Extrahepatic metastases are allowed and the primary tumor load is assessed to be intrahepatic by two or more attending physicians
   * Whether liver metastases can be resected or not is determined by two or more attending physicians according to the Chinese guidelines for the diagnosis and comprehensive treatment of colorectal liver metastases
3. Patients with unresectable colorectal liver metastases after failed standard second-line therapy

   * Including, but not limited to, Oxaliplatin, Fluorouracil, and Irinotecan
   * Treatment failure is defined as disease progression and intolerable toxicity
4. Patients who withdrew from standard therapy due to unacceptable toxicity, guaranteed to discontinue treatment before disease progression and excluded treatment with the same drug, are also allowed to be included in the study.
5. At least one measurable lesion according to RECIST 1.1 criteria
6. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
7. Subject life expectancy ≥12 weeks
8. Laboratory tests of bone marrow, hepatic and renal function and coagulation function within 7 days before the first dose of medication meet the study requirements

   - No blood transfusion, blood products, or correction with granulocyte colony-stimulating factor or other hematopoietic stimulating factor within 7 days before laboratory testing.
9. Female patients of childbearing age must have a negative blood pregnancy test within 7 days before the first dose of medication and male or female patients of childbearing age volunteered to take effective contraceptive measures during the whole treatment and within 3 months after treatment
10. All patients must sign an informed consent form and follow the trial treatment protocol and follow up plan

Exclusion Criteria:

1. ANC <1.5×109/L, or platelet count <80×109/L, or HGB < 9g/dL;

   - Blood transfusion to meet enrollment criteria within 2 weeks before enrollment is not allowed
2. serum total bilirubin>2.0 times upper limit of normal
3. AST and/or ALT>5.0 times upper limit of normal
4. Serum creatinine>1.5 times upper limit of normal, or creatinine clearance rate<50ml/min(calculated according to the Cockcroft-Gault formula)
5. APTT or PT>1.5 times upper limit of normal
6. Clinically significant severe electrolyte abnormalities by the investigator
7. Urine protein test 2+ or more, or 24 hours urine protein quantitation ≥1.0g/24h
8. Hypertension that is not stably controlled by medications: systolic blood pressure(SBP) >140mmHg or diastolic blood pressure(DBP) > 90mmHg
9. Patients with active gastric and duodenal ulcer, ulcerative colitis or other gastrointestinal diseases or unresected tumors with active bleeding, or other conditions that may cause gastrointestinal bleeding or perforation as judged by the investigators; Or patients with previous gastrointestinal perforation or gastrointestinal fistula, which is not cured after surgical treatment
10. History of arterial or deep-vein thrombosis within 6 months before enrollment or evidence or history of bleeding tendency within 2 months before enrollment, regardless of severity
11. History of troke or transient ischemic attack within 12 months before enrollment
12. History of heart disease within 6 months before enrollment, manifested as congestive heart failure, acute myocardial infarction, severe/unstable angina, coronary artery bypass grafting; impaired cardiac function in NYHA class 2 or above; left ventricular ejection fraction (LVEF) <50%
13. Uncontrolled malignant pleural, ascites, or pericardial effusion

    - defined as not being effectively controlled with diuretics or punctures
14. Clinically detectable second primary malignancy or history of other malignancies within 5 years. Adequately treated nonmelanoma skin cancers, cervical carcinoma in situ, and superficial bladder tumors [noninvasive tumors, carcinoma in situ, and T1 (tumor invasion of the lamina propria)] are excluded
15. Central nervous system (CNS) metastases or previous brain metastases
16. Clinically uncontrolled severe active infection
17. Pregnant or lactating women or women of childbearing age have a positive pregnancy test before the first dose of medication; Or female participants themselves and their partners who are unwilling to use strict contraception during the trial
18. Patients are considered by the investigator to have any clinical or laboratory abnormalities or compliance issues that precluded participation in the trial
19. Serious psychological or psychiatric abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-30 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Safety profiles by NCI-CTCAE version 5 .0 | From the first patient enrolled to 15 months after the last patient enrolled.
  The evaluation of adverse events , using NCI-CTCAE version 5.0.

SECONDARY OUTCOMES:
Overall response rate(ORR) | up to 2 years
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1.
Disease control rate(DCR) | Up to 2 years
  The ORR is defined as the proportion of subjects with confirmed complete response, partial response, or stable disease according to RECIST v 1.1.
Duration of Response (DoR) | Up to 2 years
  The time from the date of first documentation of a partial response or complete response to the date of first documentation of progressive disease (PD) or date of death due to any cause.
Response rate of intrahepatic lesions | Up to 2 years
  Response rate of intrahepatic lesions defined as the proportion of intrahepatic lesions that achieved complete response or partial response, regardless of extrahepatic lesions.
Response rate of extrahepatic lesions | Up to 2 years
  Response rate of extrahepatic lesions defined as the proportion of intrahepatic lesions that achieved complete response or partial response, regardless of intrahepatic lesions.
Quality of Life (QoL) | Up to 2 years
  The patient's ability to perform daily living can be evaluated through specific questionnaire(EORTC QLQ-C30), so as to evaluate the effect of anti-tumor drug treatment.
Overall survival (OS) | Up to 2 years
  Overall survival is defined as the time from the start of HAIC until death due to any cause.
Progression free survival (PFS) | Up to 2 years
  Progression-free survival is defined as the time from the start of HAIC until the first documentation of disease progression or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Zhu, MD, Study Chair — Peking University Cancer Hospital & Institute
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing